CLINICAL TRIAL: NCT03378297
Title: IMPACT: A Phase 0 Randomized Window-of-Opportunity Study of Novel and Repurposed Therapeutic Agents in Women Triaged to Primary Surgery for Advanced Epithelial Ovarian Cancer in Stages IIIa - IV.
Brief Title: IMPACT: A Randomized WOO Study of Novel Therapeutic Agents in Women Triaged to Primary Surgery for EOC
Acronym: IMPACT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017/1168
Record Dates: First submitted 2017-10-31; First posted 2017-12-19 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Phase 0; Window-of-opportunity; Suregry; Repurposing; Metformin; Acetylsalicylic acid; Olaparib; Letrozol
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Metformin; Aspirin; olaparib; Letrozole

STUDY DESIGN:
Intervention Model Description: The first treatment cohort has a randomized design 2:1 (olaparib 32:control 16). The study is unblinded. In the following treatment arms are initiated each will included patients (n=32) will be offered the study-prespecified treatment drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Feasibility study cohort (No Intervention)
- Metformin (Experimental): 850 mg
  Interventions: Drug: Metformin
- Acetylsalicylic acid (Experimental): 160 mg
  Interventions: Drug: Acetylsalicylic acid
- Olaparib (Experimental): 300 mg x 2
  Interventions: Drug: Olaparib
- Letrozol (Experimental): 2.5 mg
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Metformin — Metformin tablets 850 mg x 2 orally
  Arms: Metformin
Drug: Acetylsalicylic acid — Acetylsalicylic acid tablets 160 mg x1 orally
  Arms: Acetylsalicylic acid
Drug: Olaparib — Olaparib capsules 300 mg x 2 orally
  Arms: Olaparib
Drug: Letrozole — Letrozol tablets 2.5 mg x 1 orally
  Arms: Letrozol

SUMMARY:
The study will be conducted in women with advanced (stage IIIa-IV) ovarian cancer of the histologic subtype high grade serous carcinoma (HGSOC) who are going through a diagnostic laparoscopy. They will recieve treatment with a study agent for 10-14 days before surgery. They will be allocated to different study groups according to the diagnostic evaluation performed as standard of care at the department. The study is randomized and unblinded.

The primary investigational agents are:

1. Metformin tablets, 850 mg x 2 orally.
2. Acetylsalicylic acid tablets, 160 mg x1 orally
3. Olaparib capsules, 300 mg x 2 orally
4. Letrozol tablets, 2.5 mg x 1 orally

DETAILED DESCRIPTION:
The women who agree to participate in the study prior to the laparoscopic evaluation, will be allocated to different study groups according to the diagnostic evaluation performed as standard of care at the department. During inclusion in the first study cohort, the olaparib cohort (n=32), an additional 16 women are randomized as controls and will not receive neither any study drug nor placebo. The study is unblinded. There will not be randomized controls into the other study cohorts, as the control group collected will be utilized as controls for all study agents.

The women in Arm I will be included in the WOO trial, and will be treated with the study agent for 10-14 days prior to tumor reductive surgery, starting the day of laparoscopic surgery (+1 day). The treatment will be discontinued at the time of tumor reductive surgery.

Currently fourmore agents are evaluated as of particular interest, as well as feasible to introduce, in the WOO study set up: metformin, acetylsalicylic acid, olaparib, and letrozol. The first agent listed in the protocol, metformin, will be given to 32 consequtive women, and drug related analyses will thereafter be performed. The next 32 women included in the study will receive the next agent on the list, acetylsalicylic acid, while analyses for the metformin group is ongoing, and after the acetylsalicylic acid study group has been included the next agent on the list is introduced. Should any of the included women be non-eligable to receive one study drug, they will either receive the next agent on the list of the four study drugs, if eligable, or be included as control.

The women in Arm II who agree to participate in the study will not receive the study medication, but standard neoadjuvant chemotherapy until having decreased tumor load radiologically estimated and scheduled for optimal debulking procedure according to standard treatment of this group of patients. Samples from these women will be used as control in the translational part of the where we aim to identify potential molecular pathway(s) and cell type(s) that may be responsible for suboptimal debulking.

During the cancer-directed surgical procedure in participants in both Arms additional tissue samples from matching sites, preferably from tissues removed as part of the operation, as well as blood and urine samples, are obtained for comparative analysis. By use of the collected samples we can evaluate the clinical and molecular impact of the study agents among those triaged to primary cytoreductive surgery. Promising therapeutic targets identified might later be explored separately in one of the consequtive treatment study groups.

After the debulking surgery all women will follow the recommended standard of care, including chemotherapy and consolidating bevacisumab where indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a clinical diagnosis of advanced ovarian, tubal or primary peritoneal cancer. Advanced disease is defined as at least stage 3 ovarian cancer. Definition of stages will be according to the Norwegian guidelines (Norsk Gynekologisk Forening, Veileder i gynekologisk onkologi, Kapittel: Eggstokk-, tube-, bukhinnekreft. Revisjon 01.12.15). If the clinical staff in charge of the patients plan to perform cytoreductive surgery, the patient can participate in the study, irrespective of ECOG performance status. Patients must not have metastases to the central nervous system and/or carcinomatous meningitis.
2. Age 18 years or above
3. Primary treatment setting. No prior treatment for gynecological cancer. Women who have been treated surgically for cervical cancer or precancerous lesions on the cervix can be included if she has finished treatment a year or more before current diagnosis of ovarian cancer.
4. Must have laboratory values as the following :

   * White Blood Cells ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L
   * Hemoglobin ≥ 9g/dL (≥ 5.6 mmol/L)
   * Creatinine ≤ 140 μmol/L; if creatinine is borderline, the creatinine clearance ≥ 40 mL/min;
   * Bilirubin < 20 % above the upper limit of normal
   * ASAT and ALAT ≤ 2.5 the upper limit of normal
   * Albumin ≥ 2.5 g/L
   * HbA1c < 8.0 %
   * INR < 2.0
5. All laboratory tests for screening are taken maximum 14 days before start of treatment with study drug.
6. Ability to understand a written informed consent document, and the willingness to sign it.
7. Presence of adequate venous accesses for required study blood samples

Exclusion Criteria:

1. Inability to understand the information given and unable to consent and/or give the information requested, due to language, mental capacity, or disease.
2. Inability to receive substances per os.
3. Pregnancy. Pregnant women are excluded from this study, as terapeutic treatment for ovarian cancer includes teratogenic chemotherapy and surgical removal of the uterus and the ovaries.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to investigational drug or its composites.
5. History of dysregulated coagulation or known bleeding disorder.
6. Patients known to be Hepatitis B surface antigen positive, who have human immune deficiency virus (HIV) infection, and patients known or suspected to have active Hepatitis C infection.
7. Patients diagnosed or treated for other malignancy within 1 year of administration of the first dose of the study agent, or previously diagnosed with other malignancy and have residual disease. Patients with non-melanoma skin cancer or any type of carcinoma in situ will not be excluded if they have had a complete tumor resection.
8. Currently participate or have participated within the last four weeks of the first dose of the study agent in other studies including medication of participants.
9. Diagnosis of immune deficiency disorder or having received immunosuppressant treatment within the last 7 days before planned intake of the first dose of the study agent. Corticosteroids in physiologic doses can be acceptable.
10. Histologic diagnosis of non-High grade serous ovarian cancer.
11. Presence of active tumors in the central nervous system and/or carcinomatous meningitis.
12. Presence of active infection requiring systemic treatment.
13. Current diagnosis of bowel obstruction (i.e. ileus or subileus).
14. Individuals with indication of a condition, treatment or aberrant laboratory results that either can effect the results of this study or the sustainance of participation, such as renal failure stage ≥ 4, heart failure ≥ New York Heart Association (NYHA) grade III, a medical history of severe psychiatric disease, or a current diagnosis of alkoholism or drug addiction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Changes in the expression of biomarkers | 3 months
  A characterization of the tumor tissues from each patient will be performed (in pair). For each drug a specific biomarker is selected. The changes in expression of the defined biomarkers represent the primary outcome parameters. biomarkers related to the study agents and operability

CONTACTS AND LOCATIONS:
Overall Officials: Line Bjørge, MD, PhD, Principal Investigator — Helse-Bergen HF
Locations (2):
- Norway (2):
  - Helse Bergen HF, Haukeland University Hospital, Bergen
  - Helse Stavanger HF, Stavanger University Hospital, Stavanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Torkildsen CF, Austdal M, Iversen AC, Bathen TF, Giskeodegard GF, Nilsen EB, Iversen GA, Sande RK, Bjorge L, Thomsen LCV. Primary Treatment Effects for High-Grade Serous Ovarian Carcinoma Evaluated by Changes in Serum Metabolites and Lipoproteins. Metabolites. 2023 Mar 12;13(3):417. doi: 10.3390/metabo13030417. PMID 36984856
- [Derived] Torkildsen CF, Austdal M, Jarmund AH, Kleinmanns K, Lamark EK, Nilsen EB, Stefansson I, Sande RK, Iversen AC, Thomsen LCV, Bjorge L. New immune phenotypes for treatment response in high-grade serous ovarian carcinoma patients. Front Immunol. 2024 Jun 14;15:1394497. doi: 10.3389/fimmu.2024.1394497. eCollection 2024. PMID 38947323